CLINICAL TRIAL: NCT03169504
Title: Effect of Acupuncture on Patients With Chronic Obstructive Pulmonary Disease: a Multi-center, Randomized, Controlled Trial
Brief Title: Effect of Acupuncture on Patients With Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Acupuncture for COPD
Record Dates: First submitted 2017-05-21; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Acupuncture Therapy; Humans
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Acupuncture Therapy; Albuterol; Inhalation; Tiotropium Bromide; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture (Experimental): Patients in this arm will receive acupuncture.
  Interventions: Other: Acupuncture
- Conventional drug (Experimental): Patients will be individually divided into Group A, Group B, Group C and Group D according to GOLD 2017. For Group A, Salbutamol Sulphate Inhalation Aerosol (Ventolin®, GlaxoSmithKline Australia Pty Ltd) will be used. For Group B and Group C, Tiotropium Bromide Powder for Inhalation (Spiriva®, Boehringer Ingelheim International GmbH) will be used. As for Group D, Tiotropium Bromide Powder for Inhalation (Spiriva®, Boehringer Ingelheim International GmbH) or Fluticasone Propionate Powder for Inhalation (Seretide®, Laboratoire GlaxoSmithKline) will be used.
  Interventions: Drug: Conventional drug
- Acupuncture plus conventional drug (Experimental): Patients in this arm will receive both acupuncture and conventional drug.
  Interventions: Other: Acupuncture plus conventional drug

INTERVENTIONS:
Other: Acupuncture — Feishu (BL13), Dazhui (DU14) and Fengmen (BL12) will be selected as main acupoints. There are four groups of acupoints: Taiyuan (LU9) and Zusanli (ST36) for Qi deficiency of the lung ZHEGN, Taiyuan (LU9), Pishu (BL20) and Zusanli (ST36) for Qi deficiency of the lung and spleen ZHEGN, Taiyuan (LU9), Shenshu (BL23) and Zusanli (ST36) for Qi deficiency of the lung and kidney ZHEGN, and Gaohuang (BL43), Shenshu (BL23), Taixi (KI3) and Guanyuan (RN4) for Qi and Yin deficiency of the lung and kidney ZHEGN. Besides, acupoints for specific symptoms will also be considered. Hwato Sterile Acupuncture Needles For Single Use (Hwato®, Suzhou Hua Tuo Medical Instruments Co., Ltd.) size in 0.30*25 mm, 0.30*40 mm or 0.30*50 mm will be used 3 times weekly for 12 weeks.
  Arms: Acupuncture
Drug: Conventional drug — Salbutamol Sulphate Inhalation Aerosol (Ventolin®, GlaxoSmithKline Australia Pty Ltd.), 100 μg/press, 200 press, 100 μg each time (when needed), no more than 8 press daily for 12 weeks.
  Tiotropium Bromide Powder for Inhalation (Spiriva®, Boehringer Ingelheim International GmbH), 18 μg/capsule, 10 capsule, 18 μg each time, once daily for 12 weeks.
  Fluticasone Propionate Powder for Inhalation (Seretide®, Laboratoire GlaxoSmithKline), 50ug/250μg/inhalation, 60 inhalations, 50ug/250μg each time, twice daily for 12 weeks.
  Other Names: Salbutamol Sulphate Inhalation Aerosol (Ventolin®); Tiotropium Bromide Powder for Inhalation (Spiriva®); Fluticasone Propionate Powder for Inhalation (Seretide®)
  Arms: Conventional drug
Other: Acupuncture plus conventional drug — Both acupuncture and conventional drug will be used for 12 weeks treatment.
  Arms: Acupuncture plus conventional drug

SUMMARY:
This study aims to compare the efficacy of three therapies for chronic obstructive pulmonary disease (COPD) patients: one, conventional drug based on Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2017 and Chinese Medical Association Guidelines; another, acupuncture, an important part of traditional Chinese Medicine; and finally, the combination of conventional drug and acupuncture, and then determine which therapy is the most suitable for patients with COPD.

DETAILED DESCRIPTION:
COPD, characterized by progressive airflow obstruction, airway inflammation, and systemic effects or comorbidities, is a leading cause of morbidity and mortality and is projected to be the third leading cause of death worldwide by 2030. Since breathlessness, exercise limitation and health status impairment broadly exist in COPD patients, effective management should be based on an individualized assessment of disease in order to reduce both current symptoms, which involves relieving symptoms, improving exercise tolerance and health status. At present, although appropriate pharmacologic therapy can relieve COPD symptoms, reduce the frequency and severity of exacerbations, and improve health status and exercise tolerance, its cost and adverse effects can never be ignored.

Acupuncture, an important part of traditional Chinese Medicine, has been used for thousands of years in treating many painful and non-painful conditions. To date, it has become popular and widely practiced in many countries around the world. In the past two decades, acupuncture research has grown markedly, in both the proportion of randomized clinical trials (RCTs) and the impact factor of journals. Evidences from both clinicians and patients suggest that there is some beneficial effect of acupuncture on COPD.

At present, there are many therapies available for patients with COPD, it is difficult for us to identify the most suitable therapy. Thus, this study aims to compare the efficacy of conventional drug, acupuncture and the combination of conventional drug and acupuncture, and then determine which is the most suitable therapy, providing a scientific basis for clinical decision.

This is a multi-center, randomized, controlled trial to compare the efficacy of three therapies for patients with COPD. After a 14-day run-in period, 150 subjects will be randomly assigned to one of the three therapies (conventional drug, acupuncture, and the combination of conventional drug and acupuncture) for 12 weeks treatment. After the treatment period, subjects in three arms will be followed up for 12 weeks. The primary outcomes will include exercise capacity (6MWD) and St. George's Respiratory Questionnaire (SGRQ), and secondary outcomes dyspnea (mMRC), acute exacerbation, lung function, quality of life (COPD assessment test, clinical symptom assessment questionnaire, COPD-PRO and EQ-5D) and health economics.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of COPD with classification of airflow limitation severity from GOLD 1 to GLOD 3 according to GOLD 2017.
* Syndrome differentiation meets criteria of Qi deficiency of the lung ZHEGN, Qi deficiency of the lung and spleen ZHEGN, Qi deficiency of the lung and kidney ZHEGN, or Qi and Yin deficiency of the lung and kidney ZHEGN.
* Age ranges from 40 years to 80 years.

Exclusion Criteria:

* Pregnant and lactating women.
* Patients with severe cardiovascular and cerebrovascular diseases.
* Patients with severe liver and kidney disease.
* Patients with bronchiectasis, active pulmonary tuberculosis, pulmonary embolism or other severe respiratory diseases.
* Patients with tumor after resection, radiotherapy or chemotherapy in the past 5 years.
* Patients with severe neuromuscular disorders.
* Patients with severe arthritis.
* Patients with severe peripheral vascular diseases.
* Patients with severe cognitive and psychiatric disorders.
* Patients who have participated in other clinical studies in the past 4 weeks.
* Patients who have experienced one or more acute exacerbation in the past 4 weeks.
* Patients unwilling to sign informed consent.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
6MWD | Change from baseline 6MWD at week 4, week 8, week 12 of the treatment phase, and week 12 of the follow-up phase.
  6-minute walk test will be conducted to assess exercise capacity.
SGRQ | Change from baseline SGRQ score at week 12 of the treatment phase and week 12 of the follow-up phase.
  St. George's Respiratory Questionnaire (SGRQ) will be used to assess quality of life.

SECONDARY OUTCOMES:
mMRC | Change from baseline mMRC score at week 4, week 8, week 12 of the treatment phase, and week 12 of the follow-up phase.
  The modified Medical Research Council dyspnoea scale (mMRC) will be used to assess severity of dyspnea.
Frequency of acute exacerbation | Change from baseline frequency of acute exacerbation at week 4, week 8, week 12 of the treatment phase, and week 12 of the follow-up phase.
  Frequency of acute exacerbation will be recorded.
Lung function | Change from baseline lung function at week 12 of the treatment phase and week 12 of the follow-up phase.
  Spirometry will be conducted to assess lung function.
CAT | Change from baseline CAT score at week 12 of the treatment phase and week 12 of the follow-up phase.
  COPD assessment test (CAT) will be used to assess quality of life.
Clinical symptom assessment questionnaire | Change from baseline clinical symptom assessment questionnaire score at week 12 of the treatment phase and week 12 of the follow-up phase.
  Clinical symptom assessment questionnaire of COPD will be used to assess symptom.
COPD-PRO | Change from baseline COPD-PRO score at week 12 of the treatment phase and week 12 of the follow-up phase.
  COPD patient-reported outcome scale (COPD-PRO) will be used to assess quality of life.
EQ-5D | Change from baseline EQ-5D score at week 12 of the treatment phase and week 12 of the follow-up phase.
  EuroQol 5D (EQ-5D) will be used to assess quality of life.
Health economics | Up to week 12 of the follow-up phase.
  Cost of the treatment phase and follow-up phase will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Suyun Li, Professor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Li J, Xie Y, Wang Y, Wu L, Yu X, Bai L, Shao S, Zhou M, Zhang M, Yu X, Han W, Li X, Chen T. Effect of acupuncture on patients with chronic obstructive pulmonary disease: A multicenter randomized controlled trial. Complement Ther Med. 2025 May;89:103146. doi: 10.1016/j.ctim.2025.103146. Epub 2025 Feb 14. PMID 39956529